CLINICAL TRIAL: NCT05345158
Title: Robotic Retroperitoneal Lymph Node Dissection (R-RPLND) as First-line Treatment for Clinical Stage IIA/B Testicular Seminoma
Brief Title: R-RPLND as First-line Treatment for Clinical Stage IIA/B Testicular Seminoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-5242
Record Dates: First submitted 2022-03-03; First posted 2022-04-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Lymphadenopathy Retroperitoneal; Stage II Testicular Seminoma
MeSH Terms: conditions — Seminoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic Retroperitoneal Lymph Node Dissection (Experimental): Robotic retroperitoneal lymph node dissection performed using the DaVinci robotic surgical system.
  Interventions: Procedure: Robotic Retroperitoneal Lymph Node Dissection (RPLND)

INTERVENTIONS:
Procedure: Robotic Retroperitoneal Lymph Node Dissection (RPLND) — Robotic RPLND performed using the DaVinci robotic surgical system.

SUMMARY:
This study will investigate the safety and efficacy of using robotic retroperitoneal lymph node dissection (R-RPLND), a minimally invasive surgical approach, as the first-line of treatment for stage IIA/B (or equivalent) seminoma patients. R-RPLND will be trialed as an alternative to chemotherapy, radiation therapy (for seminoma patients) and open RPLND in this study.

DETAILED DESCRIPTION:
Typical treatment for testicular cancer that has spread to the retroperitoneum is chemotherapy, radiation therapy, or surgery. Chemotherapy and radiation therapy have numerous side effects and long-term complications and open retroperitoneum lymph node dissection (RPLND), the typical surgical approach for advanced testicular cancer, can be invasive and is fairly morbid. This study will investigate the safety and efficacy of using robotic retroperitoneal lymph node dissection (R-RPLND), a minimally invasive surgical approach, as the first-line of treatment for stage IIA/B (or equivalent) seminoma patients. R-RPLND will be trialed as an alternative to chemotherapy, radiation therapy (for seminoma patients) and open RPLND in this study. The primary endpoint of this study is Relapse Free Survival (RFS) at 2 years and 5 years. Secondary endpoints of this study include characteristics of relapse, time to progression, percentage of patients that can avoid chemotherapy and radiation therapy after R-RPLND, perioperative, short-term and long-term complications, rate of retrograde ejaculation, time to return of ejaculation and return to work. Additionally, Quality of Life will be measured by a questionnaire administered at 4 months post-RPLND. Approximately 25 patients will be enrolled in this study and will be followed for at least 5 years.

The data will provide important insights into the safety and efficacy of performing R-RPLND for seminoma patients with stage IIA/B (or equivalent) disease. This information will be paramount to informing clinical practice and patterns of care for treating advanced seminoma and use of the robotic approach for RPLND.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed seminomatous testicular germ cell tumour with negative margins on radical orchiectomy
* Lymphadenopathy in the retroperitoneum: at least one lymph node ≤5cm in size (in the transverse plane) detected on contrast CT scan or MRI (CS IIA/B; or active surveillance relapse with CS IIA/B equivalent)
* CT Chest negative for metastasis
* Patients qualify for this trial under the following scenarios: (1) initial diagnosis of clinical or stage IIA/B disease or (2) recurrence after surveillance for clinical stage I disease
* Patients with serum tumour marker elevation are eligible if the elevated marker does not exceed the following cut-offs within 10 days of RPLND: AFP (< 2.5 x ULN) and β-hCG (<5 IU/L)
* Curative treatment with RPLND is intended
* Under the care of a uro-oncologist at Princess Margaret Cancer Centre
* Willing to comply with follow-up protocol
* Capable of providing informed consent

Exclusion Criteria:

* Retroperitoneal lymphadenopathy >5cm in the transverse plane (CS IIC)
* Metastasis to distant lymph nodes or any organ (CS III)
* History of chemotherapy or radiotherapy to the retroperitoneum
* Patients with previous scrotal or retroperitoneal surgery for indication other than germ cell tumour
* Patients in reduced general condition, with uncontrolled intercurrent illnesses, or with life-threatening disease
* Patients with psychiatric illnesses that would limit compliance with study requirements
* Unsuitable for robotic surgery (determined by treating physician)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Relapse Free Survival (RFS) | 2 years after RPLND
  RFS is defined as the length of time between date of R-RPLND and 1) relapse or 2) death from any cause with censoring of patients lost to follow-up.
Relapse Free Survival (RFS) | 5 years after RPLND
  RFS is defined as the length of time between date of R-RPLND and 1) relapse or 2) death from any cause with censoring of patients lost to follow-up.

SECONDARY OUTCOMES:
Rate of relapse | Study duration (5 years)
  Defined as the proportion of participants experiencing relapse after primary R-RPLND. Relapse is defined as a new mass meeting size criteria (>1cm) with or without elevation of serum tumour markers.
Time to progression (TTP) | Study duration (5 years)
  TTP is defined as the time elapsed between date of R-RPLND and disease progression.
Relapse in vs. out of surgical field | Study duration (5 years)
  Relapse is classified as in vs. out of R-RPLND surgical field.
Relapse tumour characteristics | Study duration (5 years)
  Tumour size (in cm) and location
Mode of relapse detection | Study duration (5 years)
  Mode of relapse detection (e.g., CT, serum tumour markers, physical exam, etc.).
Treatment burden | Study duration (5 years)
  Number and type of treatment modalities
IGCCCG risk classification | Study duration (5 years)
  International Germ Cell Cancer Collaborative Group (IGCCCG) risk classification
Cancer-specific survival (CSS) | Study duration (5 years)
  Defined as the length of time from date of R-RPLND to the date of death from disease.
Overall survival (OS) | Study duration (5 years)
  Defined as the length of time from the date of R-RPLND until death due to any cause.
Percentage of patients that are able to avoid adjuvant treatment | Study duration (5 years)
  Percentage of patients, after treatment with R-RPLND, that are able to avoid chemotherapy and radiotherapy.
Complications | Study duration (5 years)
  Perioperative, short-term (≤30 days) and long-term (>30 days) complications. Scored using the Clavien Dindo classification system and assessed as attributable to R-RPLND by physician.
Quality of Life Surveys for Cancer Patients | 4 months post-operatively
  Measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for cancer patients (EORTC QLQ-C30).
Quality of Life Surveys for Testicular Cancer Patients | 4 months post-operatively
  Measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for testicular cancer patients (EORTC QLQ-TC26).
Return to work | Study duration (5 years)
  Self-reported by the patient and queried at each study visit until return to work.
Rate of ejaculation | Study duration (5 years)
  Self-reported by the patient and queried at each study visit until ejaculation returns.
Time of return of ejaculation | Study duration (5 years)
  Defined as the duration of time between R-RPLND and study visit when patient self-reports return of ejaculatory function.
Operative time | Duration of surgery (an average of 8 hours)
  Operative time (minutes) for surgical metrics.
Estimated blood loss | Duration of surgery (an average of 8 hours)
  Estimated blood loss (mL) for surgical metrics.
Transfusion rate | Duration of surgery (an average of 8 hours)
  Transfusion rate (mL) for surgical metrics.
Type of hemostatic agents | Duration of surgery (an average of 8 hours)
  Type of hemostatic agents used during surgery for surgical metrics.
Number of hemostatic agents | Duration of surgery (an average of 8 hours)
  Number of hemostatic agents used during surgery for surgical metrics.
Conversion rate to open surgery | Duration of surgery (an average of 8 hours)
  Conversion rate to open surgery for surgical metrics.
Number of lymph nodes resected | Duration of surgery (an average of 8 hours)
  Number of lymph nodes resected
Length of stay | Post-operatively (an average of 2 days)
  Length of stay (in days) from the date of admission to date of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hamilton, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada